CLINICAL TRIAL: NCT00969878
Title: A Double-Blind, Randomized, Placebo-Controlled, Multi-Center Study to Assess the Clinical Efficacy, Safety, and Immunogenicity of a Human Cocaine Vaccine (TA-CD) in the Treatment of Cocaine Dependence
Brief Title: Multisite Controlled Trial of Cocaine Vaccine
Acronym: TA-CD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); US Department of Veterans Affairs Cooperative Studies Program (Network); VA Maryland Health Care System (U.S. Federal Agency); Columbia University (Other); VA New York Harbor Healthcare System (U.S. Federal Agency); University of Pennsylvania (Other); Johns Hopkins University (Other); University of Cincinnati (Other); Celtic Pharma Development Services (Industry)
Responsible Party: Principal Investigator, Thomas R. Kosten, MD, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01DA025223 (NIH); R01DA025223 (NIH); DPMC (Other: NIDA); NCT00142857 (obsolete NCT alias); NCT00218088 (obsolete NCT alias)
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Cocaine Dependence
Keywords: Cocaine Vaccine, TA-CD 09
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo injection (Placebo Comparator): TA-CD placebo will be administered intra muscular. A total of 5 injections will be given over 12 weeks (i.e., at Day 1 and at the beginning of Weeks 3, 5, 9 and 13).
  Interventions: Other: Placebo Injection
- TA-CD Vaccination (Experimental): TA-CD 400 μg will be administered intramuscular. A total of 5 injections will be given over 12 weeks (i.e., at Day 1 and at the beginning of Weeks 3, 5, 9 and 13).
  Interventions: Drug: TA-CD Vaccination

INTERVENTIONS:
Drug: TA-CD Vaccination — On Day 1, subjects will be randomized to receive vaccination. Day 1 to Week 16 (3 visits per week) Subsequent vaccinations will be administered at the beginning of Weeks 3, 5, 9 and 13. There should be at least 10 days between vaccinations. Three times per week visits will be scheduled during this period through Week 16. The assessments for the active phase will be scheduled. Therapy sessions will be provided by a qualified professional such as a master's level counselor.
  Other Names: An aluminium hydroxide gel adjuvant in a saline solution.
  Arms: TA-CD Vaccination
Other: Placebo Injection — On Day 1, subjects will be randomized to receive placebo injection. Day 1 to Week 16 (3 visits per week) Subsequent placebo injections will be administered at the beginning of Weeks 3, 5, 9 and 13. There should be at least 10 days between injections. Three times per week visits will be scheduled during this period through Week 16. The assessments for the efficacy and safety monitor will be scheduled.Therapy sessions will be provided by a qualified professional such as a master's level counselor.
  Other Names: An aluminium hydroxide gel adjuvant in a saline solution.
  Arms: Placebo injection

SUMMARY:
The purpose of this study is to test the efficacy of a newly developed active vaccine against cocaine (TA-CD).

DETAILED DESCRIPTION:
This 18-week, placebo-controlled randomized clinical trial among 300 cocaine dependent patients is designed to test the efficacy of a newly developed active vaccine against cocaine (TA-CD). TA-CD vaccine consists of succinylnorcocaine (SNC) coupled to a recombinant cholera toxin B subunit (rCTB) and is designed to raise anti-cocaine antibodies in the circulation to bind to cocaine entering the bloodstream, following administration by intravenous or intranasal routes or by smoking. The antigen-antibody complexes will be too large to cross the blood-brain barrier, preventing high concentrations of cocaine reaching the brain's nucleus accumbens thereby blocking the pleasurable response to cocaine and reducing rates of drug use. The effectiveness of the vaccine is dependent on inducing sufficient levels of anti-cocaine antibodies to match the challenge from a subsequent dose of cocaine.

Because TA-CD takes several weeks to generate an antibody response, we plan to use contingency management in this interval to sustain treatment engagement. Furthermore, since TA-CD may prove most effective in patients where the antibodies can prevent a cocaine slip from turning into a binge (or return to regular use) by attenuating the priming effect, we are complementing the vaccine by using cognitive behavioral therapy (CBT) to teach patients how to cope with this priming effect and prevent a full relapse.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or female. Females either must be of non-child bearing potential (i.e., surgically sterilized or postmenopausal) or must be using adequate contraception, have a negative pregnancy test, and must agree to continue to use such precautions for 3 months after the last vaccination;
2. Meets DSM-IV-TR criteria for a principal diagnosis of cocaine dependence as confirmed by the MINI;
3. Motivated to discontinue or reduce cocaine use during the period of the study as evidenced both by the judgment of the Investigator or designee and by the subject providing at least 2 urine samples in each of the 2 baseline weeks;
4. In good general health as determined by medical history, general clinical examination, laboratory tests;
5. Has provided written informed consent. Subjects should be cooperative, willing and able to participate and adhere to the Protocol requirements.

EXCLUSION CRITERIA:

1. Subject is cocaine-free (i.e., negative urine results [BE level]) during the 2-week screening period;
2. Subject has known immunodeficiency or has a history of autoimmune disease or hypersensitivity to other vaccines. A human immunodeficiency virus (HIV) test must be performed at Screening and reported as negative for HIV-1 and HIV-2;
3. Currently taking medication known to have significant immunosuppressive effects such as systemic glucocorticoids (topical and inhaled formulations are permitted) or oral systemic corticosteroids, within 30 days prior to randomization;
4. Currently taking a dopaminergic, dopamine-blocking, dopamine-modulating, or other central dopamine-altering drug (e.g., antipsychotic drugs); a monoamine oxidase inhibitor (MAOI); or an opiate antagonist;
5. Subject has an unstable medical, neurologic, or psychiatric illness that would interfere with the subject's safety, ability to participate in the study, or the interpretability of data. Subjects who meet the DSM-IV-TR criteria for psychosis, schizophrenia, bipolar disorder or clinically significant suicidal ideation;
6. Subject had dependence on benzodiazepines, barbiturates, opiates or amphetamines according to DSM-IV-TR during the year prior to Screening. Opioid dependence includes methadone or buprenorphine maintenance treatment;
7. Subject requiring medical detox for alcohol dependence;
8. History of sensitivity to aluminium hydroxide gel;
9. History of severe adverse reaction to cholera vaccine;
10. Subject had previous vaccination with TA-CD;
11. Subject received other vaccines, including flu vaccine, within 14 days prior to signing consent;
12. Subject has participated in another clinical trial or received any other investigational compound within 14 days prior to signing consent;
13. Subject has received blood or blood products within the 3 months prior to signing consent;
14. Subject has liver function tests greater than 3 times the upper limit of normal at Screening;
15. Subject has systolic blood pressure higher than 140 mmHg and/or diastolic blood pressure >90 mmHg;
16. Female subjects with a positive pregnancy test, lactating mothers, women refusing to agree to adequate contraception and pregnancy tests during the study, or women who are planning to become pregnant during the period of the trial. Acceptable contraceptive methods are oral or parenteral hormonal contraceptives, intrauterine device (IUD), or barrier and spermicide, but not abstinence;
17. Male subjects refusing to agree to adequate contraception during the study, or males who are part of a couple planning to become pregnant during the period of the trial;
18. People who are involuntarily detained in a penal institution or people who become involuntarily detained during the study;
19. Any other factor that in the opinion of the Investigator or designee would make the subject unsafe or unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Kosten, M.D., Principal Investigator — Baylor College of Medicine
Locations (6):
- United States (6):
  - Johns Hopkins University, Baltimore, Maryland
  - NYU Langone Medical Center, New York, New York
  - Substance Abuse Treatment and Research Service (Downtown), New York, New York
  - Cincinnati Addiction Research Center, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kosten TR, Domingo CB, Shorter D, Orson F, Green C, Somoza E, Sekerka R, Levin FR, Mariani JJ, Stitzer M, Tompkins DA, Rotrosen J, Thakkar V, Smoak B, Kampman K. Vaccine for cocaine dependence: a randomized double-blind placebo-controlled efficacy trial. Drug Alcohol Depend. 2014 Jul 1;140:42-7. doi: 10.1016/j.drugalcdep.2014.04.003. Epub 2014 Apr 16. PMID 24793366
- [Derived] Martell BA, Orson FM, Poling J, Mitchell E, Rossen RD, Gardner T, Kosten TR. Cocaine vaccine for the treatment of cocaine dependence in methadone-maintained patients: a randomized, double-blind, placebo-controlled efficacy trial. Arch Gen Psychiatry. 2009 Oct;66(10):1116-23. doi: 10.1001/archgenpsychiatry.2009.128. PMID 19805702

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Injection | TA-CD Vaccination
Started | 148 | 152
Completed | 118 | 126
Not Completed | 30 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Injection | TA-CD Vaccination | Total
Number analyzed (Participants) | 148 | 152 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 148 | 152 | 300
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 38 | 72
  Male | 114 | 114 | 228
Region of Enrollment [Number; unit: participants]
  United States | 148 | 152 | 300

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Abstinence During Weeks 9 to 16 Inclusive
Description: Number of patients having at least 2 weeks of cocaine-free urines between weeks 9-16 after vaccination with five doses of TA-CD 400 µg compared to placebo
Time Frame: Over 8 weeks ( Study Weeks 9 to 16 inclusive)
Measure: Number; unit: participants
Groups:
- Placebo Injection: A saline injection to mimic the active medication is administered to the Placebo group.
- TA-CD Vaccination: The group randomized to receive the active medication, received the actual TA-CD vaccination at preset intervals as specified in the approved protocol.
Arm/Group | Placebo Injection | TA-CD Vaccination
Number analyzed (Participants) | 148 | 152
participants | 21 | 30

2. Secondary Outcome: •The Immunogenicity of TA-CD;
Description: Peak antibody levels after five vaccinations with TA-CD, which occurred at week 16.
Time Frame: During the 18 weeks study period.
Measure: Mean (95% Confidence Interval); unit: micrograms/ml
Groups:
- Placebo Injection: Subjects randomized to the placebo group were injected with a saline solution on the same schedule as those in the active medication group.
- TA-CD Vaccination: Subjects randomized to the active medication group were injected with the active TA-CD at preset intervals per protocol specifications.
Arm/Group | Placebo Injection | TA-CD Vaccination
Number analyzed (Participants) | 118 | 126
micrograms/ml | 0 [0 to 0] | 59 [0 to 186]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo Injection | TA-CD Vaccination
Serious Adverse Events (participants affected / at risk) | 15/148 | 14/152
Other Adverse Events (participants affected / at risk) | 0/148 | 0/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Injection (N=148) | TA-CD Vaccination (N=152)
Depression with suicidality (Psychiatric disorders) | 6 (6) | 5 (5)
Other hospitalizations (General disorders) | 9 (9) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No